CLINICAL TRIAL: NCT04779723
Title: Comparison of Laparoscopic Sleeve Gastrectomy (LSG) With Laparoscopic Gastric Bypass (LRYGB) in Bariatric Surgery; 30-Days Post-Operative Complications in Bariatric Surgery
Brief Title: 30-Days Post-Operative Complications in Bariatric Surgery
Acronym: Bariatric
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Multan Medical And Dental College (Other)
Responsible Party: Principal Investigator, Manzar Ali, Consultant General and laparoscopic Surgeon, Multan Medical And Dental College
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: MMDC-2018-023
Record Dates: First submitted 2021-02-07; First posted 2021-03-03 (Actual); Last update posted 2021-03-03 (Actual); Status verified 2021-02

CONDITIONS: Bariatric Surgery
Keywords: Bariatric surgery; Laparoscopic Roux-en-Y gastric bypass; Laparoscopic sleeve gastrectomy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- LRYGB Procedure (Active Comparator): LRYGB technique was performed by placing 4 to 6 trocars, a 150 cm ante-colic Roux-limb gastric pouch (30 to 50 ml) was created with linear stapled or circular stapled gastro-jejunostomy, a 50-cm long biliopancreatic limb was chosen. A passive drainage was kept near to the gastro-jejunostomy.
  Interventions: Procedure: Comparison of two Techniques of bariatric surgery
- LSG Procedure (Active Comparator): 35 Fr bougie was used for the calibration of a gastric tube. 3 to 6 cm of longitudinal incision of the stomach was done at pylorus to the angle of His. Using of absorbable suture, the staple line was sewn.
  Interventions: Procedure: Comparison of two Techniques of bariatric surgery

INTERVENTIONS:
Procedure: Comparison of two Techniques of bariatric surgery — We compared the 30 days outcomes in patients who underwent LSG procedure with those who underwent LRYGB

SUMMARY:
comparison of 30-days post-operative outcomes of laparoscopic sleeve gastrectomy (LSG) and laparoscopic Roux-en-Y gastric bypass (LRYGB)

DETAILED DESCRIPTION:
Obesity is one of the most challenging chronic diseases in the western world as well as in Pakistan. Half of the people in this world consider themselves overweight or obese. Obesity is one of the most challenging chronic diseases in the western world as well as in Pakistan . Half of the people in this world consider themselves overweight or obese. Obesity is challenging to control by medical therapy and drug treatment. The most effective way to treat obesity is bariatric surgery. Laparoscopic Roux-en-Y gastric bypass (LRYGB) is a "gold standard" bariatric surgical procedure. Recently there is much attention gained by laparoscopic sleeve gastrectomy (LSG). Therefore, we decided to conduct this comparative study to compare the early post-op complications of LSG with LRYGB technique in patients undergoing bariatric surgery.

ELIGIBILITY:
Inclusion Criteria:

* patients of age 18 to 65 years
* body mass index (BMI) >35 kg/m2 (Morbidly obese)
* Patients with failed conservative treatment of weight control

Exclusion Criteria:

* Severe indicative gastroesophageal reflux disease (GERD)
* Conversion of another bariatric procedure
* Large hiatal hernia
* Patients with inflammatory bowel disease

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 116 (Actual)
Dates: Start 2018-06-13 (Actual); Primary Completion 2019-02-12 (Actual); Study Completion 2019-10-12 (Actual)

PRIMARY OUTCOMES:
Frequency of Anastomotic Leakage in Each Study Arm | within the first 30 days after surgery
  Patients were examined on postoperative 30 days for the presence of Anastomotic leakage
Frequency of Bleeding in Each Study Arm | 24 hours after surgery
  Patients were examined postoperative for the presence of bleeding
Number of Infections in Each Study Arm | 30 days
  Patients were examined on postoperative 30 days for the presence of Wound infections
Mortality in Each Study Arm | 30 days
  Patients were followed for 30 days and number of mortalities was noted on each arm

SECONDARY OUTCOMES:
Hospital Stay | 30 days
  Duration of hospitalization

CONTACTS AND LOCATIONS:
Locations (1):
- Multan Medical and Dental College, Multan, Punjab Province, Pakistan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Gallagher EJ, LeRoith D, Karnieli E. The metabolic syndrome--from insulin resistance to obesity and diabetes. Endocrinol Metab Clin North Am. 2008 Sep;37(3):559-79, vii. doi: 10.1016/j.ecl.2008.05.002. PMID 18775352
- [Background] Chooi YC, Ding C, Magkos F. The epidemiology of obesity. Metabolism. 2019 Mar;92:6-10. doi: 10.1016/j.metabol.2018.09.005. Epub 2018 Sep 22. PMID 30253139
- [Background] Siddiqui M, Hameed R, Nadeem M, Mohammad T, Simbak N, Latif A, et al. Obesity in Pakistan; current and future perceptions. J Curr Trends Biomed Eng Biosci. 2018;17:001-004
- [Background] Adams TD, Davidson LE, Litwin SE, Kolotkin RL, LaMonte MJ, Pendleton RC, Strong MB, Vinik R, Wanner NA, Hopkins PN, Gress RE, Walker JM, Cloward TV, Nuttall RT, Hammoud A, Greenwood JL, Crosby RD, McKinlay R, Simper SC, Smith SC, Hunt SC. Health benefits of gastric bypass surgery after 6 years. JAMA. 2012 Sep 19;308(11):1122-31. doi: 10.1001/2012.jama.11164. PMID 22990271
- [Background] Suter M, Donadini A, Romy S, Demartines N, Giusti V. Laparoscopic Roux-en-Y gastric bypass: significant long-term weight loss, improvement of obesity-related comorbidities and quality of life. Ann Surg. 2011 Aug;254(2):267-73. doi: 10.1097/SLA.0b013e3182263b66. PMID 21772127
- [Background] Li K, Gao F, Xue H, Jiang Q, Wang Y, Shen Q, Tian Y, Yang Y. Comparative study on laparoscopic sleeve gastrectomy and laparoscopic gastric bypass for treatment of morbid obesity patients. Hepatogastroenterology. 2014 Mar-Apr;61(130):319-22. PMID 24901132
- [Background] Peterli R, Borbely Y, Kern B, Gass M, Peters T, Thurnheer M, Schultes B, Laederach K, Bueter M, Schiesser M. Early results of the Swiss Multicentre Bypass or Sleeve Study (SM-BOSS): a prospective randomized trial comparing laparoscopic sleeve gastrectomy and Roux-en-Y gastric bypass. Ann Surg. 2013 Nov;258(5):690-4; discussion 695. doi: 10.1097/SLA.0b013e3182a67426. PMID 23989054